CLINICAL TRIAL: NCT06283654
Title: Relieving the Emergency Department by Using a 1-lead ECG Device for Atrial Fibrillation Patients After Pulmonary Vein Isolation: a Historically Controlled Prospective Trial
Brief Title: Relieving the Emergency Department by Using a 1-lead ECG Device for Atrial Fibrillation Patients After Pulmonary Vein Isolation
Acronym: relievED
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Luuk Hopman, prof dr, Amsterdam UMC, location VUmc
Other Study IDs: VUmc 2018.539
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Atrial Fibrillation
Keywords: 1-lead ECG; ED visits
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1-lead ECG group: Patients after PVI that received a 1-lead ECG
  Interventions: Device: 1-lead ECG
- standard care group: standard care group

INTERVENTIONS:
Device: 1-lead ECG — patient were handed out a 1 lead ECG device, they were free to use it anyway they wanted, even not at all
  Groups: 1-lead ECG group

SUMMARY:
In this study, the researchers explored a new approach to manage atrial fibrillation, a disease that affects millions worldwide. The goal was to see if using a simple handheld ECG device for monitoring heart rhythm could help patients avoid unnecessary visits to the emergency department (ED) after undergoing a common procedure known as pulmonary vein isolation (PVI). This procedure is often used to treat AF, but following it patients frequently visit the ED due to concerns about their heart rhythm, which can strain healthcare resources. The researchers proved a group of patients with a 1-lead ECG device , which allowed users to check their heart rhythm at any time. The researchers compared the ED utilization over a year with that of patients who received standard care after PVI. The hope was that by using the 1-lead ECG device, patients could better manage their condition from home and only seek medical help when truly necessary.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a prevalent and clinically significant cardiac arrhythmia, with a growing incidence. The primary objectives in AF management are symptom relief, stroke risk reduction, and prevention of tachycardia-induced cardiomyopathy. Two key strategies for rhythm control include antiarrhythmic drug therapy and pulmonary vein isolation (PVI), with PVI being recommended for selected patients. Even though PVI is effective, post procedural health care utilization is high, contributing to emergency department (ED) overcrowding, which is a global healthcare concern. The use of remote rhythm diagnostics, such as a 1-lead ECG device, may mitigate this issue by reducing ED visits and facilitating more plannable AF care. Objective: This study aimed to assess whether providing AF patients with a 1-lead ECG device for 1 year after PVI would reduce ED utilization compared to standard care. Additionally, the study assessed whether this would enhance plannability of AF related healthcare utilization. Methods: A historically controlled, prospective clinical trial was conducted. The 'intervention' group are patients undergoing PVI for AF, all patients in this group receive a KM device for 1 year for remote rhythm monitoring. The historical control group were patients undergoing PVI between January 2016 and December 2017; these patients did not receive a KM. Data on ED visits, planned and unplanned cardioversions, and outpatient contacts in the year after the PVI were collected for both groups.

ELIGIBILITY:
Inclusion Criteria:

* AF and PVI

Exclusion Criteria:

* <18y

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with all kinds of AF who underwent a PVI
Sampling Method: Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
number of ED visits | 1 year after PVI

SECONDARY OUTCOMES:
ratio of the number of cardioversions emergency vs planned | 1 year after PVI

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC -vumc, Amsterdam, Netherlands

REFERENCES:
- [Derived] Selder JL, Mulder MJ, van de Vijver WR, Croon PM, Wentrup LE, van der Pas SL, Twisk JWR, Tulevski II, Van Rossum AC, Allaart CP. Does providing atrial fibrillation patients, after pulmonary vein isolation, with a 1-lead ECG device relieve the emergency department?-A historically controlled prospective trial. PLOS Digit Health. 2024 Dec 20;3(12):e0000688. doi: 10.1371/journal.pdig.0000688. eCollection 2024 Dec. PMID 39705212